CLINICAL TRIAL: NCT02784925
Title: Evaluate Patients With Chronic Hepatitis Before and After Treatment of Body Index by Three-dimensional Force-controlled Ultrasound Measurement of Subcutaneous Fat
Brief Title: Evaluate Patients With Chronic Hepatitis by Three-dimensional Force-controlled Ultrasound Measurement
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Taipei Medical University WanFang Hospital (Other)
Collaborators: Taipei Medical University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: N201603045
Record Dates: First submitted 2016-05-20; First posted 2016-05-27 (Estimated); Results first posted 2017-06-22 (Actual); Last update posted 2017-06-22 (Actual); Status verified 2016-04

CONDITIONS: Fatty Liver
MeSH Terms: conditions — Fatty Liver | interventions — Ultrasonography

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- fatty liver subjects (Other): Ultrasound (US) B mode image is an alternative method to measure tissue structure and has proven to be an accurate technique to measure subcutaneous fat thickness.
  Interventions: Device: Ultrasound (US) B mode image

INTERVENTIONS:
Device: Ultrasound (US) B mode image — Ultrasound (US) B mode image is an alternative method to measure tissue structure
  and has proven to be an accurate technique to measure subcutaneous fat thickness.

SUMMARY:
Ultrasound (US) B mode image is an alternative method to measure tissue structure and has proven to be an accurate technique to measure subcutaneous fat thickness. However, pressing the transducer onto the skin with too much force will significantly reduce the subcutaneous adipose tissue thickness. In this study, a force controlled system combined with US transducer was used for 3D subcutaneous fat imaging and reconstruction.

DETAILED DESCRIPTION:
The diagnosis of fatty liver (steatosis) is made when fat in the liver exceeds 5-10% by weight. Fatty liver (FL) is commonly associated with alcohol or metabolic syndrome (diabetes, hypertension, obesity, and dyslipidemia), but can also be due to any one of many causes. Most people were detected from serum lipid abnormalities in the physical examination, and confirmed as the fatty liver disease by ultrasound imaging. In some previous studies, ultrasound was reported to provide an accurate and reliable measurement tool for the thickness measurements of subcutaneous adipose tissue. This method can overcome some limitations of the skinfold thickness measurements. Ultrasound (US) B mode image is an alternative method to measure tissue structure and has proven to be an accurate technique to measure subcutaneous fat thickness. However, pressing the transducer onto the skin with too much force will significantly reduce the subcutaneous adipose tissue thickness. In this study, a force controlled system combined with US transducer was used for 3D subcutaneous fat imaging and reconstruction. Finally, the correlations between body fat percentage and subcutaneous fat in steatosis patients have been investigated. The body fat percentage was determined by dual energy X-ray absorptiometry (DEXA, GE Lunar iDXA canner) and bioelectrical impedance analysis (BIA, Omron，HBF-370), and then, the correlation between body fat percentage and subcutaneous adipose tissue in normal and steatosis patients have been evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 20-65 adults who are confirmed have fatty liver by echo

Exclusion Criteria:

* none

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2016-06; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Fatty Liver Subjects: Ultrasound (US) B mode image is an alternative method to measure tissue structure and has proven to be an accurate technique to measure subcutaneous fat thickness.
  Ultrasound (US) B mode image: Ultrasound (US) B mode image is an alternative method to measure tissue structure
  and has proven to be an accurate technique to measure subcutaneous fat thickness.
Period: Overall Study
Arm/Group | Fatty Liver Subjects
Started | 30
Completed | 30
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Fatty Liver Subjects
Number analyzed (Participants) | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 30
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21
  Male | 9

OUTCOME MEASURES:

1. Primary Outcome: Subcutaneous Fat in Steatosis Patients
Time Frame: up to 6 months
Population: fatty liver patients
Measure: Mean (95% Confidence Interval); unit: cm^3
Arm/Group | Fatty Liver Subjects
Number analyzed (Participants) | 30
cm^3
  female__abdomen | 9.54 [6.79 to 13.98]
  male__abdomen | 10.48 [4.65 to 16.81]
  female__front thigh | 5.24 [3.34 to 11.60]
  male__front thigh | 4.09 [1.89 to 9.12]

ADVERSE EVENTS:
Groups:
- Fatty Liver Subjects: Ultrasound (US) B mode image is an alternative method to measure tissue structure and has proven to be an accurate technique to measure subcutaneous fat thickness.Ultrasound (US) B mode image: Ultrasound (US) B mode image is an alternative method to measure tissue structure and has proven to be an accurate technique to measure subcutaneous fat thickness.
Arm/Group | Fatty Liver Subjects
Serious Adverse Events (participants affected / at risk) | 30/30
Other Adverse Events (participants affected / at risk) | 30/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Fatty Liver Subjects (N=30)
fatty liver (Hepatobiliary disorders) | 30 (30)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Fatty Liver Subjects (N=30)
refuse to have body measurement (Social circumstances) | 30 (30)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes